CLINICAL TRIAL: NCT01993355
Title: A Multidisciplinary Approach to Treat and Rehabilitate Patients With Chronic Low Back Pain
Brief Title: Chronic Low Back Pain: A Multidisciplinary Approach
Acronym: CLBP-HUVH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CLBP-PT_ATR_274-2012
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Pain
Keywords: non-specific chronic low back pain,; health-related quality of life,; physioterapy,; sophrology,; cognitive-behavioral therapy,; motivational interviewing
MeSH Terms: conditions — Chronic Pain | interventions — Physical Therapy Modalities; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAU (Active Comparator): Control group. Treatment as usual (TAU): Physiotherapy program for CLBP.
  Interventions: Other: Physiotherapy
- Intervention 1 Relaxation techniques-sophrology (Experimental): Intervention group 1: TAU + relaxation techniques-sophrology program.
  Interventions: Other: Physiotherapy; Other: Intervention 1
- Intervention 2 Cognitive-behavioral therapy (Experimental): Intervention group 2: TAU + cognitive-behavioral therapy.
  Interventions: Other: Physiotherapy; Behavioral: Intervention 2

INTERVENTIONS:
Other: Physiotherapy — Physical therapy exercise program for CLBP patients. Its goal is to reduce pain and improve patients' health-related quality of life, functional capacity and well-being.
  Other Names: Treatment as usual (TAU)
Other: Intervention 1 — Relaxation techniques-sophrology consists of a set of physical and relaxation exercises that include breathing methods, visualization, modification of states of consciousness, etc. with the goal to enhance balance between body and mind to improve health-related quality of life, reduce pain and foster patients' well-being.
  Other Names: Relaxation techniques-sophrology
  Arms: Intervention 1 Relaxation techniques-sophrology
Behavioral: Intervention 2 — Cognitive-behavioral therapy (in combination with motivational interviewing principles) is aimed to facilitate psychological adjustment and self-management of CLBP with the ultimate goal of increasing patients' health-related quality of life and well-being.
  Other Names: CBT
  Arms: Intervention 2 Cognitive-behavioral therapy

SUMMARY:
Introduction: Non-specific chronic low back pain (CLBP) is one of the most frequent causes for patient disability and a general recurrent cause for medical consultation with high costs to public health. From rehabilitative medicine, physiotherapy is commonly offered. Although this treatment is aimed to reduce disability, pain severity and pain-related anxiety-depressive symptoms, many patients report partial improvement and recurrent intensive and disabling pain episodes. Therefore, a new approach in the treatment and rehabilitation of this pathology that takes into account psychosocial aspects that might be modulating pain is necessary.

Material and methods: This project aims to assess the efficacy of two complementary interventions to standard physical therapy, such as relaxation techniques and cognitive-behavioral intervention, to improve health-related quality of life (HRQoL) among patients with CLBP. It is hypothesized that groups receiving these complementary interventions will significantly improve their adherence to physiotherapy and the control of their pain and, ultimately, these aspects will facilitate a decreasing of pain intensity and better HRQoL.

For these purposes, a pre-post longitudinal design will be carried out, with follow-up assessments at 6 and 12 months in a sample of 66 participants. This sample will be divided into: control group (physiotherapy), intervention group 1 (physiotherapy and relaxation techniques-sophrology) and intervention group 2 (physiotherapy and cognitive-behavioral intervention).

Expected impact: Study results are not available yet. However, if working hypotheses are confirmed, a multidisciplinary model of care for CLBP will be empirically justified. This approach is expected to benefit HRQoL among these patients implying a significant short-mid term reduction of public health costs.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific chronic (> 6 months of evolution) low back pain diagnosis
* Ability to read and speak in Spanish

Exclusion Criteria:

* Addictive behaviors (DAST-10 > 3, alcoholism, drug addiction or other drug abuse)
* Psychiatric contraindications (BDI > 15 or other severe psychiatric disorder not stabilized)
* Neurological impairment
* No mental competence (MEC < 23)
* Fibromyalgia and/or chronic fatigue

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The SF-12v2 Health Status Questionnaire (change is being assessed) | Baseline, 6 and 12 months
  The SF-12 measures health-related quality of life including items from various domains both physical and psychological.

SECONDARY OUTCOMES:
VAS for Self-perceived Pain | Baseline, 6 and 12 months
  Visual Analogue Scale to rate self-perceived pain. Recall period: last 4 weeks.
Oswestry-15 Disability Index | Baseline, 6 and 12 months
  The Oswestry Disability Index (aka: Oswestry Low Back Pain Disability Questionnaire) is a time-tested outcome assessment tool that is used to measure a patient's impairment and quality of life (i.e., how badly the pain has affected their life).

OTHER OUTCOMES:
LISAT-8 | Baseline, 6 and 12 months
  The LISAT is a domain-specific measure of life satisfaction, which corresponds to Box E (subjective evaluations and reactions; life satisfaction) of Dijker's Model.
STAI | Baseline, 6 and 12 months
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to screen anxiety and to distinguish it from depressive syndromes.
BDI-13 | Baseline, 6 and 12 months
  The Beck Depression Inventory (BDI) is a 13-item (short-form), self-report rating inventory that measures characteristic attitudes and symptoms of depression.
PSQI | Baseline, 6 and 12 months
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality during the previous month.
CAD | Baseline and 12 months
  The CAD (Cuestionario para el Afrontamiento al Dolor) is a coping questionnaire to chronic pain developed in a Spanish sample.
TAS-20 | Baseline and 12 months
  The Toronto Alexithymia Scale (TAS) 20-item is one of the most commonly used measures of alexithymia (people who have trouble identifying and describing emotions and who tend to minimise emotional experience and focus attention externally).
PSS-14 | Baseline and 12 months
  The Perceived Stress Scale (PSS) is a 14-item questionnaire that measures the degree to which life events are considered stressful.
DUKE-11 | Baseline and 12 months
  The DUKE 11-item social support questionnaire measures an individual's perception of the amount and type of personal social support. The original instrument included 14 items, grouped into 4 subscales: Quantity of Support, Confidant Support, Affective Support, and Instrumental Support.
VAS for patient satisfaction with treatment received | Baseline, 6 and 12 months
  Visual Analogue Scale to rate patients' satisfaction with treatment, attention received and outcomes.
Medical and demographics | Baseline
  Medical (medical and psychopathological history, physical exploration of LBP and possible substance abuse or other toxic habits such as alcohol or tobacco) and demographics (age, gender, immediate family network, education, job and SES) of patients are collected according to standard procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Carmina Castellano-Tejedor, PhD, Principal Investigator — Hospital Universitari Vall d'Hebron - Institut de Recerca Vall d'Hebron; Elisa Barnola-Serra, MD, Study Director — Hospital Vall d'Hebron; Gemma Costa-Requena, MsC, Study Chair — Hospital Vall d'Hebron; Pilar Lusilla-Palacios, MD, PhD, Study Chair — Hospital Vall d'Hebron; Alex Ginés-Puertas, Study Chair — Hospital Universitario Vall d'Hebron - Parc Sanitari Pere i Virgili; Laura Camprubí-Roca, Study Chair — Hospital Universitario Vall d'Hebron - Parc Sanitari Pere i Virgili; Mª Lluisa Torrent-Bertran, MD, Study Chair — Hospital Vall d'Hebron; Ana Palacios-González, Study Chair — Hospital Universitario Vall d'Hebron - Parc Sanitari Pere i Virgili; Tamara Biedermann-Villagra, MD, Study Chair — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari Vall d'Hebron Institut de Recerca Vall d'Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Group of pain for patients with chronic low back pain: A multidisciplinary intervention. Lusilla-Palacios, P, Castellano-Tejedor, C, Barnola-Serra, E, Ramos-Rondón, C, Biedermann-Villagra, T, Torrent-Bertran, M.L, Costa-Requena, G, Camprubí-Roca, L, Palacios-González, A, Cuxart-Fina, A, Ginés-Puertas, A, Bosch-Graupera, A. Poster communication on the 21th European Congress of Psychiatry, Nice, France, 25-29/05/2010.
- [Result] Castellano-Tejedor, C., Costa-Requena, G., Lusilla-Palacios, P., Biedermann-Villagra, T., Barnola-Serra, E. Calidad del sueño en pacientes con lumbalgia crónica inespecífica. Rehabilitación 48(4): 219-225, 2014. DOI: 10.1016/j.rh.2014.05.003
- [Result] Castellano-Tejedor, C., Costa-Requena, G., Lusilla-Palacios, P., Barnola-Serra, E. Calidad de vida en pacientes con dolor lumbar crónico: efectos de un programa de intervención multidisciplinar a los 6 meses de seguimiento. Comunicació tipus pòster presentada a les II Jornades BiblioPro del Parc de Recerca Biomédica de Barcelona, Barcelona 19 de febrer de 2015.